CLINICAL TRIAL: NCT06485440
Title: The Effects of Preoperative Botulinum Toxin A Injection Prior to Abdominal Wall Reconstruction Procedures on Respiratory System Function
Brief Title: The Effects of Preoperative Botulinum Toxin A Injection on Respiratory System Function
Status: Completed | Type: Observational
Sponsor: Swissmed Hospital (Other)
Responsible Party: Principal Investigator, Mateusz Zamkowski, Principal Investigator, Director, Swissmed Hospital
Other Study IDs: BTA Impact
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Botulinum Toxins, Type A; Hernia
Keywords: BTA; Hernia; AWR; Loss of Domain; Prehabilitation; Incisional; Botulinum Toxin A
MeSH Terms: conditions — Hernia; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BTA: 10 patients with giant hernias of the anterior abdominal wall (W3 in the classification of the European Hernia Society) prepared with BTA injections prior to surgery
  Interventions: Drug: Dysport 300 UNT Injection

INTERVENTIONS:
Drug: Dysport 300 UNT Injection — 300 UNITS of BTA (Dysport) injected to lateral abdominal muscles prior to abdominal wall reconstruction (4 weeks before surgery)
  Other Names: BTA Injections

SUMMARY:
Hernias are common complications post-abdominal surgeries, often leading to significant issues such as "loss of domain," where organs shift permanently, reducing abdominal cavity capacity. This complicates surgeries as there is insufficient space to reposition organs. A growing method to address this involves preoperative botulinum toxin A (BTA) injections into lateral abdominal muscles. BTA induces temporary paralysis, expanding the abdominal cavity and aiding muscle approximation for hernia repair. Initiated in 2009, this approach is particularly used for defects over 10cm. However, standardized protocols are lacking, and the impact on respiratory function remains under-researched. This study aims to evaluate the effects of preoperative BTA injections on respiratory volumes. Ten patients will undergo pulmonary function tests before and after BTA injections. The study will focus on changes in respiratory efficiency, given the respiratory challenges associated with large hernias and the "loss of domain" effect.

DETAILED DESCRIPTION:
Hernias are frequent complications following abdominal procedures, particularly in cases of large defects which may lead to the "loss of domain" effect. This phenomenon involves permanent displacement of organs into an alternative space, reducing the effective capacity of the peritoneal cavity. Surgical management of giant hernial sacs is challenging due to insufficient space within the abdominal cavity to accommodate organ repositioning.

Abdominal wall reconstruction specialists have developed various techniques to address these complexities. One increasingly utilized method involves the injection of botulinum toxin A (BTA) into the lateral abdominal muscles (external oblique, internal oblique, and transverse muscles). BTA induces temporary muscular paralysis lasting approximately 6-8 months. This paralysis extends the muscle compartment, thereby increasing abdominal cavity volume. This expansion facilitates the approximation of rectus abdominis muscles and the closure of fascial defects.

Initial attempts to employ BTA for the treatment of giant abdominal hernias began in 2009. Since then, its role in abdominal wall surgery has grown steadily. Optimal timing for surgery post-BTA injection is typically 3-4 weeks, when maximal muscle extension and abdominal volume increase (up to 20-30%) are observed.

Despite widespread clinical use, standardized protocols for BTA application remain lacking due to limited comparative studies and small sample sizes in existing literature. Rare allergic reactions aside, comprehensive documentation of adverse effects from BTA injections remains minimal. However, variability in patient response suggests potential differences in treatment efficacy.

Respiratory efficiency poses a significant challenge in patients with giant abdominal hernias, exacerbated by the "loss of domain" effect which impairs diaphragm function and alters respiratory mechanics. Predicting perioperative outcomes is further complicated by advanced age, comorbidities, and obesity among affected patients.

To investigate the impact of preoperative BTA injection on respiratory function, a study will assess pulmonary volumes using spirometry in 10 patients with giant hernias of the anterior abdominal wall (classified as W3 by the European Hernia Society). Participants will undergo spirometry before and 4 weeks after lateral muscle group BTA injection as part of preoperative evaluation for abdominal wall reconstruction at the Swissmed Hospital Hernia Centre in Gdansk.

The injection of BTA will be performed in outpatient settings, under ultrasound guidance. Each patient received 300 units of BTA (Dysport®, IPSEN, Boulogne-Billancourt, France), with 150 units administered to each side. The BTA administration procedure will begin with drawing lines on the skin to mark the lower edge of the last rib and the upper edge of the iliac crest. Then, a line connecting both marked sections is drawn along the anterior axillary line. On this line, three equally spaced points will be marked. These will be the sites for needle insertion and BTA administration. 300 units of BTA will be dissolved in 150ml of 0.9% saline. This solution will be then divided into six 25ml portions. Each portion is administered at the previously designated points. During the injection at a point, under ultrasound control, we reach the transverse muscle and administer 8ml of the solution. Then, the needle will be withdrawn to the internal oblique muscle, and another 8ml is administered. Finally, the needle will be withdrawn to the level of the external oblique muscle, where the remaining portion of the dose is administered. This procedure is repeated at each point

ELIGIBILITY:
Inclusion Criteria:

1. Large abdominal hernia (at least W3 in the EHS classification), requiring additional preoperative techniques to prevent ACS (abdominal compartment syndrome) in the postoperative period.
2. Age >18 years.
3. Written consent to participate in the study.
4. Health status allowing the safe conduct of surgery.

Exclusion Criteria:

1. Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with giant hernias of the anterior abdominal wall (W3 in the classification of the European Hernia Society) will be included in this study. Patients qualified for the reconstruction of the anterior abdominal wall, qualified by an expert team from the Hernia Centre (Swissmed Hospital in Gdansk) and meeting the inclusion criteria for the study. Each patient, as part of preoperative preparation, will have pulmonary function tests performed twice, i.e., spirometry, before and 4 weeks after injecting the lateral muscle groups with BTA.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
FVC (forced vital capacity) | 4-6 weeks
  FVC before and 4-6 after BTA injection
FEV1 (forced expiratory volume in one second) | 4-6 weeks
  FEV1 before and 4-6 after BTA injection
PEF (peak expiratory flow) | 4-6 weeks
  PEF before and 4-6 after BTA injection

OTHER OUTCOMES:
MEF (Maximal Mid Expiratory Flow) | 4-6 weeks
  MEF before and 4-6 after BTA injection
FIVC (Forced Inspiratory Vital Capacity) | 4-6 weeks
  FIVC before and 4-6 after BTA injection

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Śmietański, MD, PhD, Prof., Study Director — Swissmed Hospital; Mateusz Zamkowski, MD, PhD, Study Chair — Swissmed Hospital
Locations (1):
- Swissmed Hospital, Gdansk, Gdańsk, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on justified cases.

REFERENCES:
- [Result] Elstner KE, Jacombs AS, Read JW, Rodriguez O, Edye M, Cosman PH, Dardano AN, Zea A, Boesel T, Mikami DJ, Craft C, Ibrahim N. Laparoscopic repair of complex ventral hernia facilitated by pre-operative chemical component relaxation using Botulinum Toxin A. Hernia. 2016 Apr;20(2):209-19. doi: 10.1007/s10029-016-1478-6. Epub 2016 Mar 7. PMID 26951247
- [Result] Timmer AS, Claessen JJM, Atema JJ, Rutten MVH, Hompes R, Boermeester MA. A systematic review and meta-analysis of technical aspects and clinical outcomes of botulinum toxin prior to abdominal wall reconstruction. Hernia. 2021 Dec;25(6):1413-1425. doi: 10.1007/s10029-021-02499-1. Epub 2021 Sep 21. PMID 34546475
- [Result] Weissler JM, Lanni MA, Tecce MG, Carney MJ, Shubinets V, Fischer JP. Chemical component separation: a systematic review and meta-analysis of botulinum toxin for management of ventral hernia. J Plast Surg Hand Surg. 2017 Oct;51(5):366-374. doi: 10.1080/2000656X.2017.1285783. Epub 2017 Feb 20. PMID 28277071
- [Result] Whitehead-Clarke T, Windsor A. The Use of Botulinum Toxin in Complex Hernia Surgery: Achieving a Sense of Closure. Front Surg. 2021 Oct 1;8:753889. doi: 10.3389/fsurg.2021.753889. eCollection 2021. PMID 34660688
- [Result] Zendejas B, Khasawneh MA, Srvantstyan B, Jenkins DH, Schiller HJ, Zielinski MD. Outcomes of chemical component paralysis using botulinum toxin for incisional hernia repairs. World J Surg. 2013 Dec;37(12):2830-7. doi: 10.1007/s00268-013-2211-6. PMID 24081529
- [Result] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905